CLINICAL TRIAL: NCT00281138
Title: Pediatric Asthma Disparities: Perceptions and Management
Brief Title: Center for Reducing Asthma Disparities - Rhode Island/Puerto Rico Centers
Status: Completed | Type: Observational
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1197; U01HL072438 (NIH)
Record Dates: First submitted 2006-01-20; First posted 2006-01-24 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2008-07

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
To reduce disparities in asthma among Latino children.

DETAILED DESCRIPTION:
BACKGROUND:

Asthma is a serious chronic condition affecting over 14 million Americans, but the prevalence rates are higher in certain populations (e.g. 10 percent in inner-cities and 30 percent among the homeless vs. 5 percent in a general population of whites). African Americans and Hispanics from the Northeast are twice as likely to die from asthma as whites. African Americans are four times as likely to be hospitalized for asthma and are five times more likely than whites to seek care for asthma at an emergency department. Reasons for these higher rates are not certain, and most likely result from an interaction of risk factors such as environmental exposures, genetic predisposition, access to appropriate medical care, socioeconomic status, and cultural health practices. The National Heart, Lung, and Blood Institute supports a variety of activities to address the pressing public health problems posed by asthma. However, progress in reducing disparities has been disappointingly slow. Separate, independent research projects have generated important clues for understanding the nature and scope of the problem. A more coordinated, interdisciplinary and comprehensive approach to research is needed to take advantage of these clues, move the science further and faster, and increase our capacity to improve health outcomes among minority and economically disadvantaged populations. Cooperative centers of research that foster partnerships among minority medical centers, research intensive institutions, and the communities in which asthma patients live will promote such advancement.

The Request for Applications for the Centers for Reducing Asthma Disparities was released in October, 2001. The objective of the program is to promote partnerships (called Centers) between a minority serving institution (MSI) that may not have a strong research program and a research intensive institution (RII) that has a track record of NIH-supported research and patient care. The purpose of the partnership is to conduct collaborative research on asthma disparities (i.e. greater prevalence of asthma, higher rates of morbidity due to asthma, and lesser access or use of quality medical care among minorities and poor).

DESIGN NARRATIVE:

The Rhode Island : Puerto Rico Asthma Center (RIPRAC) has been established to reduce disparities in asthma among Latino children. Brown University faculty involved with an extensive pediatric asthma research program will join with epidemiologists, clinicians, and health services researchers from the minority serving University of Puerto Rico to study potentially overlooked determinants of disparity. A training component (based on a successful T32 research training program) will involve individuals from both sites at both sites. The Rhode Island : Puerto Rico Asthma Center includes four projects that seek to understand the causes of disparities at multiple levels : the biomedical, the individual/family, and the socioenvironmental level. The four projects, respectively, will 1) examine discrepancies between the diagnosis of asthma as assessed by parental report, the primary care medical record and our systematic diagnosis based on the NHLBI guidelines; 2) assess characteristics (prescription practices, shared decision making, continuity and access to care) of the health care system that may differentially affect asthma morbidity; 3) evaluate family beliefs, the burden of asthma management and medication adherence as they affect asthma morbidity and health care utilization in Latino and Anglo children; and 4) study the relation of symptom perception to pediatric asthma discrepancies. Subjects for all four projects will be the same 300 mainland Anglos, 200 mainland Latinos (of Puerto Rican and Dominican descent) and 400 island Puerto Rico children with asthma, aged 7-15, thereby promoting comparability and efficiency. Chi-square analyses and ANOVA's will be used to assess differences between groups; techniques of logistic regression and multiple regression will be used to model the effects of covariates. The Center Training component will provide clinical research education and supervision to Puerto Rican trainees and faculty, enhance cultural awareness of Brown personnel as it relates to asthma disparities, and launch at least three trainee-led pilot research projects in the area.

ELIGIBILITY:
1) Diagnosed asthma or history of breathing problems (coughing, wheezing, shortness of breath) in the 12 months prior to study enrollment; 2) Non-Latino white, Puerto Rican or Dominican ethnic background; 3)ages 7-15 years

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with asthma or a history of breathing problems, from Non-Latino white, Puerto Rican or Dominican ethnicities. Participant recruitment occurred in Rhode Island and in island Puerto Rico.
Sampling Method: Non-Probability Sample
Enrollment: 983 (Actual)
Dates: Start 2002-09; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Asthma morbidity | 12 months retrospective and 3 months prospective

CONTACTS AND LOCATIONS:
Overall Officials: Glorisa Canino, Principal Investigator — University of Puerto Rico; Gregory Fritz, Principal Investigator — Rhode Island Hospital